CLINICAL TRIAL: NCT03546062
Title: Lipid Accumulation in Heart Transplant From Non-diabetic Donors to Diabetic Recipients
Brief Title: Diabetes and Lipid Accumulationand Heart Transplant
Acronym: DCM-AHEAD
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Raffaele Marfella, primary investigator, University of Campania Luigi Vanvitelli
Other Study IDs: DCM-AHEAD
Record Dates: First submitted 2018-05-22; First posted 2018-06-06 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus; Heart Failure
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The patients received in the past heart transplant. In the removed and frizzed hearts authors will extract portions of septal wall. From this tissue authors will analyze inflammatory markers and microRNAs involved in the progression of cardiac disease.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- T2DM patients treated by HTx: Authors will include a population of T2DM patients with advanced heart failure and treated by heart transplant. 41 patients recluted from January 2015
  Interventions: Other: patients treated by HTx
- T2DM Metformin treated by HTx: Authors will include a population of T2DM patients with advanced heart failure and treated by heart transplant in metformin therapy. 35 patients recluted from January 2015
  Interventions: Other: patients treated by HTx
- Non-diabetic patients treated by HTx: Authors will include a population of non-diabetic patients with advanced heart failure treated by heart transplant. 82 patients recluted from January 2015
  Interventions: Other: patients treated by HTx

INTERVENTIONS:
Other: patients treated by HTx — From removed and frozen hearts, authors will conduct a tissue and molecular analysis of possible mechanisms T2DM linked.

SUMMARY:
Idiopathic dilated cardiomyopathy (IDC) is defined by the presence of left ventricular systolic dysfunction in the absence of an abnormal loading condition or significant coronary artery disease. IDC is the main cause of end-stage heart failure (HF) and is responsible for half of all heart transplants (HTx). Endocrine disorders, including diabetes, are known to be associated with IDC. Diabetes mellitus (DM), which is present in 75% of patients with idiopathic IDC, is an independent risk factor for the development of heart failure and death in IDC. Therefore, DM can exacerbate the need for HTx, in addition, diabetic patients are less suitable for HTx and DM remains an independent risk factor for death even after HTx. Recent studies have revealed the presence of diabetic cardiomyopathy, a condition of myocardial dysfunction without coronary artery disease. This term was introduced for the first time by Rubler et al. in 1972 which highlighted patients with diabetes and congestive heart failure with normal coronary arteries. The pathophysiological mechanisms through which diabetes affects the development and progression of diabetic heart disease are not known. Therefore, the purpose of our study will be to evaluate, in the explanted diabetic heart, the presence of possible cellular alterations attributable to the diabetic disease. Furthermore, the progression of these lesions in the transplanted heart in diabetic patients will be evaluated.

DETAILED DESCRIPTION:
BACKGROUND Heart failure (HF) is an increasing disease, with a prevalence and incidence of about 1% and 0.15% of the general population respectively, affecting at least 300,000 patients in the USA. However, in cases of advanced heart failure, refractory to maximal medical therapy, and to devices supporting the heart rhythm and cardio-circulatory function, the only valid therapeutic option remains the cardiac transplant. Diabetic patients with advanced heart failure seem to benefit from this therapy not differently as compared to non-diabetics. On other hand, in patients with advanced heart failure and selected for heart transplantation, the diabetes may condition a different degree of structural and molecular pathology that is not present, or present at least in a different way in non-diabetics selected for same HF etiology, clinical features, and HF stage. Therefore, in this study authors will study the anatomical-pathological, cellular, and molecular characteristics, as the pathways of inflammatory, oxidative, apoptotic and epigenetic expression in diabetics vs. non diabetics affected by idiopathic dilated cardiomyopathy (IDCM) and therefore in the absence of ischemic heart disease, and referred to Heart Center for cardiac transplantation. Authors' study hypothesis is that diabetes can condition a different degree of structural, cellular, and molecular pathology in patients with IDCM Vs. non-diabetic patients, due to excessive metabolic activity, with increased synthesis and release of inflammatory, oxidative, and apoptotic molecules. These investigations will be focused on microscopic, histological and functional analysis of the cellular metabolism of cardiac tissue extracted from diabetics vs. non diabetics IDCM patients, and removed during cardiac transplantation. However, in a subsequent ex vivo phase authors will evaluate cellular, molecular, inflammatory and epigenetic effectors related to the different microscopic tissue pattern obtained from myocardial tissue samples. From authors' investigations, these new identified targets of the HF molecular and cellular processes in diabetics vs. non diabetics, may be used in the future as specific therapeutic targets to improve clinical outcomes in IDCM diabetics with advanced heart failure.

MATERIALS AND METHODS Study population Authors will enroll a population of IDCM diabetics and non diabetics selected to receive a heart transplant. This study will be conducted at the Department of Medical Sciences, at the Department of Cardiac Surgery, and at the Department of Biochemistry of the University of Campania "Luigi Vanvitelli". Selection, randomization and enrollment of patients will be carried out at the Department of Medical Sciences, followed by clinical follow up; Cardiac transplantation and cardiac tissue sampling will be performed at the Cardiosurgery Department; Molecular and cellular studies will be conducted at the biochemistry department. The follow-up will be 12 months. The diabetic pathology will be diagnosed according to the international guidelines of the American Heart Association.

Inclusion criteria: patients aged > 18, <75 years, with indication to receive a heart transplant (survival score for accepted heart failure accepted (HFSS) at high risk, peak VO2 <10 ml / kg / min after reaching the anaerobic threshold; arrhythmias recurrent symptomatic ventricles refractory to medical treatment, ICD and surgical), affected by IDCM with heart failure in NYHA class III / IV refractory to maximal medical therapy; diabetic and non-diabetic patients Exclusion criteria: contraindication to receiving cardiac transplantation; non-idiopathic dilated cardiopathy (valvulopathies, ischemic-infarct cardiopathy, etc.), acute myocardial infarction, acute heart failure, neoplastic disease, and chronic diseases that may influence the inflammatory profile both systemic and cardiac (cancer, chronic intestinal inflammation, hepatitis, AIDS) , and a life expectancy <6 months. All patients will be included in the study after signing informed consent to participate in the study. Routine analysis will be performed upon enrollment in the study, before cardiac transplantation and follow-up. During the follow-up (figure 1) clinical examinations, routine ecg and echocardiography will be performed regularly. Molecular study and cell study will be performed on myocardial tissue from explanted hearts. The study will be performed according to the Helsinki declaration.

Intervention In this observational study, authors will evaluate a cohort of consecutive patients (diabetic vs. non-diabetic) affected by IDCM and heart failure in class III / IV NYHA refractory to maximal medical therapy and treated at the Division of Cardiac Surgery of the University of Campania "Luigi Vanvitelli "by cardiac transplantation. The study will be conducted in three different parts: human study, ex vivo cell study, molecular study.

Human study: conducted in the Department of Medical Sciences and Cardiac Surgery, the enrolled patient will be treated by heart transplant, according to the international guidelines governing cardiac transplantation. After cardiac transplantation, a biopsy of myocardial tissue of the removed heart will be performed. The intervention will be conducted at the Cardiosurgery Division of the "Luigi Vanvitelli" University of Campania.

Cardiac tissue analysis A portion of muscle tissue (50 grams) will be removed from the explanted heart, from which 3 portions will be obtained: a portion will be incorporated in the OCT compound and frozen in liquid nitrogen for immunohistochemical analysis, a second portion will be immediately frozen in nitrogen liquid and stored at -70 ° C for the isolation of RNA, and a third portion will be weighed, cut into small pieces (2 mm3) and transferred to a 12-well plate. Based on the weight of the tissue, serum-free DMEM (2 ml / g) will be added to the well and incubated at 37 ° C in a mild-fluctuated CO2 incubator. At 3 hours, the conditioned soils will be collected and centrifuged at 4 ° C for 10 minutes. The supernatants from cultures of epiphonic and subcutaneous adipose tissue will be stored in aliquots at -70 ° C for the measurement of inflammation mediators released by ELISA.

Blood samples

Blood collection will be carried out on the morning of surgery and during the follow-up phases by peripheral venous blood taken in tubes without pyrogen with or without EDTA as anticoagulant. For plasma, the EDTA tubes will be placed on melted ice, then centrifuged within 20 minutes at 1500 g for 10 minutes at 4 ° C. The plasma will be stored in aliquots at 80 ° C for all ELISA tests. Serum glucose, lipid panels and inflammatory markers will be analyzed in the University of Campania's Biochemistry Laboratory.

Inflammatory markers

The authors will analyze the mediators of plasma and cardiac inflammation with ELISA (R & D systems) according to the procedure recommended by the manufacturer. ELISA standard kit they will be used for IL-6 measurements, and highly sensitive ELISA kits for TNF-alpha and IL-1 measurements. Intra-assay variability will be set at 10%, while inter-assay variability will be 15%.

RNA analysis and Real-Time Reverse Transcription

Samples of myocardial tissue will be minced in a TriZol reagent (Invitrogen) and homogenized completely on ice. The total RNA will be extracted from the chloroform and purified twice through the mini RNAasy columns. After the DNase treatment on a column, the RNA will be eluted with RNase-free water. Transcripts encoding various inflammatory mediators will be measured by the TaqMan real-time reverse-polymerase-RT (PCR) chain reaction with the TaqMan Gold RT-PCR and the PRISM 7700 Sequence Detection System (Applied Biosystems). PCR primers and TaqMan probes will be obtained from Applied Biosystems and optimized according to the manufacturer's protocol. The PCR reaction conditions will be at 48 ° C for 30 minutes, at 95 ° C for 10 minutes, followed by 40 cycles of 95 ° C for 15 seconds and 60 ° C for 1 minute. The GAPDH transcripts will be amplified in a separate tube to normalize the variance in the input RNA. The mRNA in various samples will be estimated by the relative standard method with a series of dilutions of RNA from human vascular cells or from leukocytes.

Immunohistochemistry The authors will obtain frozen sections (10 m), which will be air-dried for 15 minutes and immersed in xylene for 10 minutes to remove the fat. The sections will then be hydrated in decreasing degrees of alcohol and stained with hematoxylin and eosin. The selected serial sections will be immunosimochemical with the Universal Elite ABC (Vector Laboratories) kit according to the manufacturer's protocol. Briefly, the sections will be incubated with 0.3% H2O2 in methanol for 30 minutes, followed by a block with horse serum or 5% goat. After washing in PBS, the sections will be incubated with primary antibodies for 1 hour in a wet chamber. Subsequently, the slides will be incubated with secondary antibodies for 30 minutes followed by avidin-biotin for 30 minutes. The sections will then be exposed to DAB and counterstained with hematoxylin. The following antibodies will be used: CD3 (Tlymphocyte, 1:50, Novocastra), CD68 (monocytes / macrophages, 1: 100, Dako) and triptases (mast cells, 1:50, Novocastra).

Follow-up After being discharged from the hospital, all patients will be required to carry out control visits, as indicated by the authors on the management of patients post-transplant cardiac, at the Division of Cardiac Surgery of the University of Campania "Luigi Vanvitelli "and the sixth division of Internal Medicine of the University of Campania" Luigi Vanvitelli ". All patients will be monitored for 12 months after follow-up, by clinical evaluation (ECG, stress test, echocardiogram) to maintain HbA1c levels <7%, fasting glycemia between 90 and 140 mg / dl and post-prandial glycemia <180 mg / dl, as indicated in the guidelines for the management of diabetic and post-CABG patients. In the 12 months of follow-up, patient management will be conducted by telephone interview, physical examination (at discharge and 3, 6 and 12 after cardiac transplantation), ecg and echocardiography (at discharge and 3, 6 and 12 after cardiac transplantation); CMRI will be conducted at baseline and 12 months after CABG. Similarly, the bio-humoral evaluation will be conducted during all the follow-up phases.

Statistical Analysis The study population groups (diabetics vs. non-diabetics) will be compared using the Pearson test for categorical variables and the Kruskal-Wallis test for continuous variables. Candidates for admission to the multivariate model will be identified by focusing on factors that will differ significantly (P value <0.05) in the univariate analysis between diabetics vs. non-diabetics. Cox regression will be used to construct the predictive model of mortality. The risk ratio for mortality will be adjusted for age, BMI, cholesterol, LDL, triglycerides and aspirin, ticlopidine, anti-aggregating agents, beta-blockers, ACE inhibitors or sartans, antidiabetic drugs, statins, etc. present at the time of hospitalization for cardiac transplantation. Analysis of survival after cardiac transplantation will be performed using the Kaplan-Meier curve and Cox regression method. Mortality curves will be obtained separately for diabetic patients compared to non-diabetic patients, and then compared using the log-rank test. All tests will be considered significant if with a value of p <0.05. All analyzes will be conducted in 2 populations: diabetic vs non-diabetic patients after cardiac transplantation. For all analyzes the SPSS program will be used (version 21, IBM SPSS).

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus (T2DM);
* heart failure in III/IV NYHA class
* patients with clear indication to receive heart transplantation (HTx).

Exclusion Criteria:

* aged < 18 years
* aged >75 years
* non T2DM diagnosis
* controindication to receive HTx.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two main groups according to whether patients did or did not have pre-transplantation diabetes. Patients with DM for at least 6 months before HTX, with optimal glycemic control (HbA1c <7.0), BMI <30kg/m2, without severe secondary end-organ disease will be included. Patients with endomyocardial biopsy specimens consistent with ISHLT Grade 2R considered positive for rejection, increased T4/T8 ratio, positive IgM and/or IgG Cytomegalovirus antibodies, and with post-HTX diabetes will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Marfella, MD, Principal Investigator — Università della Campania Luigi Vanvitelli
Locations (2):
- Italy (2):
  - Celestino Sardu, Naples
  - Raffaele Marfella, Naples

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marfella R, D'Onofrio N, Mansueto G, Grimaldi V, Trotta MC, Sardu C, Sasso FC, Scisciola L, Amarelli C, Esposito S, D'Amico M, Golino P, De Feo M, Signoriello G, Paolisso P, Gallinoro E, Vanderheyden M, Maiello C, Balestrieri ML, Barbato E, Napoli C, Paolisso G. Glycated ACE2 reduces anti-remodeling effects of renin-angiotensin system inhibition in human diabetic hearts. Cardiovasc Diabetol. 2022 Aug 5;21(1):146. doi: 10.1186/s12933-022-01573-x. PMID 35932065
- [Derived] Marfella R, D'Onofrio N, Trotta MC, Sardu C, Scisciola L, Amarelli C, Balestrieri ML, Grimaldi V, Mansueto G, Esposito S, D'Amico M, Golino P, Signoriello G, De Feo M, Maiello C, Napoli C, Paolisso G. Sodium/glucose cotransporter 2 (SGLT2) inhibitors improve cardiac function by reducing JunD expression in human diabetic hearts. Metabolism. 2022 Feb;127:154936. doi: 10.1016/j.metabol.2021.154936. Epub 2021 Nov 18. PMID 34801581
- [Derived] Marfella R, Amarelli C, Cacciatore F, Balestrieri ML, Mansueto G, D'Onofrio N, Esposito S, Mattucci I, Salerno G, De Feo M, D'Amico M, Golino P, Maiello C, Paolisso G, Napoli C. Lipid Accumulation in Hearts Transplanted From Nondiabetic Donors to Diabetic Recipients. J Am Coll Cardiol. 2020 Mar 24;75(11):1249-1262. doi: 10.1016/j.jacc.2020.01.018. PMID 32192650

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetic Group With Metformin Therapy: Patients with DM for at least 6 months before HTX, with optimal glycemic control (HbA1c <7.0), and metformin therapy without severe secondary end-organ disease (retinopathy, neuropathy or nephropathy) were included
- Diabetic Group Without Metformin Therapy: Patients with DM for at least 6 months before HTX, with optimal glycemic control (HbA1c <7.0), without metformin therapy and severe secondary end-organ disease (retinopathy, neuropathy or nephropathy) were included
- Non-diabetic Group: Patients without DM for at least 6 months before HTX, with optimal glycemic control (HbA1c <7.0), without end-organ disease (retinopathy, neuropathy or nephropathy) were included
Period: Overall Study
Arm/Group | Diabetic Group With Metformin Therapy | Diabetic Group Without Metformin Therapy | Non-diabetic Group
Started | 41 | 46 | 90
Completed | 35 | 41 | 82
Not Completed | 6 | 5 | 8
Not completed — Adverse Event | 6 | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Diabetic Group Without Metformin Therapy: Authors will include a population of T2DM patients with advanced heart failure and treated by heart transplant. 41 patients recluted from January 2015
  patients treated by HTx: From removed and frozen hearts, authors will conduct a tissue and molecular analysis of possible mechanisms T2DM linked.
- Diabetic Group With Metformin Therapy: Authors will include a population of T2DM patients with advanced heart failure and treated by heart transplant in metformin therapy. 35 patients recluted from January 2015
  patients treated by HTx: From removed and frozen hearts, authors will conduct a tissue and molecular analysis of possible mechanisms T2DM linked.
- Non-diabetic Patients: Authors will include a population of non-diabetic patients with advanced heart failure treated by heart transplant. 82 patients recluted from January 2015
  patients treated by HTx: From removed and frozen hearts, authors will conduct a tissue and molecular analysis of possible mechanisms T2DM linked.
- Total: Total of all reporting groups
Arm/Group | Diabetic Group Without Metformin Therapy | Diabetic Group With Metformin Therapy | Non-diabetic Patients | Total
Number analyzed (Participants) | 41 | 35 | 82 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (5.6) | 50 (6.6) | 52 (5.5) | 51 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  SEX: Female | 11 | 9 | 22 | 42
  SEX: Male | 30 | 26 | 60 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 41 | 35 | 82 | 158
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 41 | 35 | 82 | 158
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 41 | 35 | 82 | 158
ejection fraction [Mean (Standard Deviation); unit: percent] | 35 (3) | 37 (2) | 36 (4) | 36 (3)

OUTCOME MEASURES:

1. Primary Outcome: Myocyte Lipid Accumulation as Oil Red-O Positive Biopsie
Description: Authors will evaluate myocyte lipid accumulation as Oil Red-O positive biopsie after heart transplant at follow up.
Time Frame: 12 months.
Population: myocyte lipid accumulation as Oil Red-O positive biopsies
Measure: Count of Units; unit: Endomyocardial Biopsies
Units Other Than Participants: Endomyocardial Biopsies
Groups:
- Diabetic Metformin Group: Patients with DM for at least 6 months before HTX, with optimal glycemic control (HbA1c <7.0), treated with metformin without severe secondary end-organ disease (retinopathy, neuropathy or nephropathy) were included
- Diabetic Group Without Metformin Therapy: Patients with DM for at least 6 months before HXT, with optimal glycemic control, that were not treated with metformin.
- Non-diabetic Group: Patients without diabetes
Arm/Group | Diabetic Metformin Group | Diabetic Group Without Metformin Therapy | Non-diabetic Group
Number analyzed (Participants) | 35 | 41 | 82
Number analyzed (Endomyocardial Biopsies) | 105 | 123 | 246
Endomyocardial Biopsies | 54 | 21 | 0

ADVERSE EVENTS:
Time Frame: 12 month
Description: heart rejection
Groups:
- Diabetic Without Metformin Group: Patients with DM for at least 6 months before HTX, with optimal glycemic control (HbA1c <7.0), that were not treated with metformin, without severe secondary end-organ disease (retinopathy, neuropathy or nephropathy) were included
- Non Diabetic Patients: Patients without diabetes
Arm/Group | Diabetic Metformin Group | Diabetic Without Metformin Group | Non Diabetic Patients
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/41 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/41 | 0/82
Other Adverse Events (participants affected / at risk) | 0/35 | 0/41 | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetic Metformin Group (N=35) | Diabetic Without Metformin Group (N=41) | Non Diabetic Patients (N=82)
rejection (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Our real life study is not multi-center study and thus we need to extend our observations to a larger cohort of randomized patients. Second, immunosuppressive therapy by per se could affect molecular mechanisms of DMCM.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT03546062/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT03546062/ICF_001.pdf